CLINICAL TRIAL: NCT04316234
Title: Acute Health Effects of Passive Exposure to Particles From Electronic Cigarettes - a Randomized Controlled Double-blinded Cross-over Trial Among COPD Patients
Brief Title: Acute Health Effects of Passive Vape Among COPD Patients
Acronym: PASVAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Torben Sigsgaard, Professor, Doctor, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1711000
Record Dates: First submitted 2020-02-05; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Electronic Cigarette Use; Second Hand Smoke; Lung Function
Keywords: Electronic cigarettes; Secondhand vape; Health effects; Lung function; Biomarkers; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Vaping; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: A randomised double-blinded cross-over study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Vaping was done in another chamber and thereby led into the exposure chamber, so it could not be observed. On days with clean air, vapers were chewing nicotine gum instead of vaping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A. Clean Air (No Intervention): Clean air - no vaping was done.
- B. Passive vaping (Experimental): E-cigarette users were present in an adjacent chamber during both exposures, but only in situation B they were vaping and the vape-polluted air was passed on to the exposure chamber.
  Interventions: Other: Passive vape

INTERVENTIONS:
Other: Passive vape — On days with passive vape, 2-3 vapers in an adjacent chamber were vaping by turn, and vape was passed on to the exposure chamber continuously .
  Arms: B. Passive vaping

SUMMARY:
The use of e-cigarettes is often permitted in otherwise smoke-free areas causing passive vape exposure for present individuals. Little is known about the potential adverse health effects of passive vape, and people with respiratory diseases may be more susceptible.

The aim of the present study was to investigate local and systemic effects of short-term passive exposure to vape from e-cigarettes among patients with mild or moderate chronic obstructive pulmonary disease COPD in a randomized controlled double-blinded cross-over study.

DETAILED DESCRIPTION:
Introduction: The use of e-cigarettes is often permitted in otherwise smoke-free areas causing passive vape exposure for present individuals. Little is known about the potential adverse health effects of passive vape, and people with respiratory diseases may be more susceptible.

Aim: to investigate local and systemic effects of short-term passive exposure to vape from e-cigarettes among patients with mild or moderate chronic obstructive pulmonary disease (COPD).

Design: In a randomised double-blinded cross-over study non-smoking COPD patients were exposed for four hours at two different exposure conditions separated by 14 days; A) clean filtered air and B) passive vaping under controlled environmental conditions.

Measurements: TSI P-TRAK Ultrafine Particle Counter was used for particle counts. Health effects, including lung function (FEV1/FVC) and fraction of exhaled nitric oxide (FeNO) were evaluated in relation to local and systemic effects prior to, right after and 24 h. after exposure.

Analysis: Mixed methods approach taking both time and exposure into account.

ELIGIBILITY:
Inclusion Criteria:

* Never smoker or ex-smokers ≥ 6 months
* Aged 18+
* A known diagnosis of COPD (FEV1/FVC < lower limit of normal, app. 70%)
* MRC ≥ 2 or CAT score ≥ 10

Exclusion Criteria:

* Exposure to smoking more than 30 min./day
* Treatment with inhaled or oral corticosteroids
* Known hypersensitivity to constituents in e-cigarettes
* Any other disease that could influence the study parameters
* Conditions that prevent safe access to the climate chambers (such as claustrophobia)
* Perennial rhinitis
* Deformed nasal airways
* Not being able to change from long-acting medication to short-acting medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Particles in Exhaled Air (Surfactant Protein A & Albumin) | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  PExA: Subjects performed repeated breath maneuvers allowing for airway closure and re-opening, and exhaled particles were optically counted and collected on a membrane using the (novel) PExA® instrument set-up.

SECONDARY OUTCOMES:
Change in Lung Function (FEV1 & FVC) | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  Spirometry
Change in Fractional exhaled nitric oxide (FENO) | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  NIOX system; Aerocrine AB, Sweden
Change in Blood samples | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  IL-8, Nightingale analyses for biomarkers
Change in nasal volume (using Acoustic rhinometry) | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  Is used to assess the nasal cross sectional area and volume. The left and right nasal cavity were studied alternatively until three reproducible measurements were obtained. The minimum cross sectional cavity area was calculated from the means of the measurements. By integration of the area-distance curve, the sum of the volume 2 to 4 (vol2-4) from the nostril was determined on both sides.
Change in Symptom questionnaire | Every 30 min during 4 hours of exposure.
  In the exposure chamber participants were asked to fill out a symptom questionnaire every 30 min. regarding their well-being and experienced symptoms in eyes, nose and mouth.
Change in biomarkers in Saliva Sample | At baseline (0 hour), after exposure (4 hours), and the day after exposure (24 hours)
  An oral svap from Salivette was placed in the mouth of the participant to collect saliva by gently chewing the swab for one minute. Afterwards the saturated swab was removed to the suspended insert and closed firmly with a lid. Then the sample was transferred to a freezer and stored for -80 C until further analysis. The sample will be analyzed for biomarkers (amylase, cortisol, substance P, lysozyme and secretory IgA.)

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Laursen, MSc, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Central Region Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No